CLINICAL TRIAL: NCT03342157
Title: Pilot Study for the Efficacy and Tolerability of Senokot-S in the Treatment of Diabetic Gastroparesis
Brief Title: Docusate/Senna for the Treatment of Diabetic Gastroparesis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17.120
Record Dates: First submitted 2017-11-10; First posted 2017-11-14 (Actual); Results first posted 2020-10-23 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Gastroparesis
MeSH Terms: interventions — doxidan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High-dose (Experimental): 8.6/50 mg of senna/docusate, oral, twice daily
  Interventions: Drug: senna/docusate
- Low-dose (Experimental): 8.6/50 mg of senna/docusate, oral, once daily
  Interventions: Drug: senna/docusate

INTERVENTIONS:
Drug: senna/docusate — Stimulant laxative
  Other Names: Senokot-S

SUMMARY:
The aim of the study is to evaluate the efficacy of the stimulant laxative Senokot-S® for the treatment of diabetic gastroparesis. Senokot-S, and its metabolites, are thought to produce peristalsis, drive intraluminal fluid and electrolyte shifts, and have an irritant effect on the gut mucosa. These complex physiologic mechanisms appear may sufficiently promote stomach emp-tying, and thereby reduce or eliminate the severity of gastroparesis symptoms. In this open label study, participants will be randomized into high and low dose groups to assess for ideal dosing and tolerability. It is the overall goal of this study to select the most promising dose-strength for the treatment of mild through severe gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, male and non-pregnant, non-lactating females
* Diagnosis of type 1 or type 2 diabetes mellitus
* Clinical diagnosis of diabetic gastroparesis

Exclusion Criteria:

* Diagnosed idiopathic gastroparesis
* A history or inflammatory bowel disease, such as Crohn's disease or ulcerative colitis
* A history of bowel obstruction, current unexplained abdominal pain, or undiagnosed rectal bleeding
* Gastrointestinal cancer
* Any active cancer
* Prior gastric surgery
* End-stage heart disease, liver disease, lung disease
* Known or suspected drug abuse
* Any condition requiring use of daily narcotics
* Concurrent usage of mineral oil or products containing mineral oil
* Current or recent (within the last 3 months) usage of Senokot-S, docusate or senna

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Gose, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Health Care, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from 11/01/2017 through 05/11/2020 at St Lukes Medical Center utilizing outpatient and inpatient referrals from practitioners.
Pre-assignment Details: No enrolled participants were excluded from the study.
Period: Overall Study
Arm/Group | High-dose | Low-dose
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-dose | Low-dose | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 51 [51 to 51] | 49 [49 to 49] | 50 [49 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2
modified gastroparesis cardinal symptom index daily diary (mGCSI-DD) [Number; unit: participants] — Statistical analysis not appropriate on a sample size of 1. Population: Statistical analysis not appropriate on a sample size of 1.
breakthrough medication use [Number; unit: participants] — Statistical analysis not appropriate on a sample size of 1. Population: Statistical analysis not appropriate on a sample size of 1.
frequency of bowel habits [Number; unit: participants] — Statistical analysis not appropriate on a sample size of 1. Population: Statistical analysis not appropriate on a sample size of 1.

OUTCOME MEASURES:

1. Primary Outcome: Modified Gastroparesis Cardinal Symptom Index-Daily Diary (mGCSI-DD)
Description: mGCSI-DD uses 6-point Likert scale from 0 (none) to very severe (5)
Time Frame: 28 days
Population: Statistical analysis not appropriate on a sample size of 1 patient per arm.
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Frequency of Use of Breakthrough Medication
Description: Change in the frequency of use of breakthrough medication - daily diary
Time Frame: 28 days
Population: Statistical analysis not appropriate on a sample size of 1 patient per arm.
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Frequency of Bowel Movements
Description: Change in the frequency of bowel movements - daily diary
Time Frame: 28 days
Population: Statistical analysis not appropriate on a sample size of 1 patient per arm.
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | High-dose | Low-dose
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
study stopped due to low enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT03342157/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03342157/ICF_001.pdf